CLINICAL TRIAL: NCT05549453
Title: Use of Nexstim SNBT System in Its Intended Use
Brief Title: Use of Nexstim SNBT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nexstim Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NX140344
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Usability of the Graphical User Interface of the Device for Its Intended Use

STUDY DESIGN:
Intervention Model Description: The purpose of the investigation is to assess the usability of the new device user interface in a feasibility study conducted with a prototype device utilizing the new interface in an open label use of the device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- SNBT device use (Experimental): SNBT device is used for motor cortex localization, motor threshold determination and for targeting the intracranial electric field induced by the device to the intarcranial location required for the use of the device for its intended use
  Interventions: Device: Nexstim SNBT use

INTERVENTIONS:
Device: Nexstim SNBT use — Active device use

SUMMARY:
The clinical investigation assesses the usability of the new graphical user interface of the Nexstim SNBT device in its intended clinical uses. The hardware and the technical functionality of the device of the SNBT device are in other respects similar to those of the earlier Nexstim NBT device, which has been cleared by FDA for treatment of Major Depressive Disorder in 2017 (K170902) and has received EU CE mark for the same and for treatment of chronic neuropathic pain.

The present investigation is not intended to establish the safety and efficacy of the SNBT device. Rather, the purpose is to assess the usability of the new user interface in a feasibility study conducted with a prototype device utilizing the new user interface.

ELIGIBILITY:
Inclusion Criteria:

* age 18-64 years signed informed consent form

Exclusion Criteria:

* pregnant implanted electrical device ferromagnetic metal anywhere in the body metal in head except amalgam dental fillings epilepsy migraine previous head trauma or surgery a diagnosed neurological disorder medication affecting the central nervous system

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of usability of the graphical user interface for use of the device in its intended use | Up to 3 months. From subject's enrollment to end of subject's study participation.
  yes/no assessment by an expert clinical user of the technology

SECONDARY OUTCOMES:
Assessment of usability of the graphical user interface for use for motor cortex localization by device use | Up to 3 months. From subject's enrollment to end of subject's study participation.
  yes/no assessment by an expert clinical user of the technology
Assessment of usability of the graphical user interface for use for motor threshold determination by device use | Up to 3 months. From subject's enrollment to end of subject's study participation.
  yes/no assessment by an expert clinical user of the technology
Assessment of usability of the graphical user interface for the targeting of the intracranial electric field generated by the device to the intracranial target location required for the use of the device in its intended use | Up to 3 months. From subject's enrollment to end of subject's study participation.
  yes/no assessment by an expert clinical user of the technology
Assessment of whether the usability of the graphical user interface is superior to that experienced by the user during his/her previous experience with earlier NBT product generations | Up to 3 months. From subject's enrollment to end of subject's study participation.
  yes/no assessment by an expert clinical user of the technology

CONTACTS AND LOCATIONS:
Overall Officials: Jarmo T Laine, MD,PhD, Principal Investigator — Nexstim Ltd
Locations (1):
- Nexstim Plc, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No